CLINICAL TRIAL: NCT01474499
Title: A Multi-center, Randomized, Single-blind Clinical Study of the Comparative Safety and Efficacy of Docusate Sodium and Sorbitol Rectal Solution and Glycerine Enemas in Patients With Constipation
Brief Title: A Trial of Docusate Sodium and Sorbitol Rectal Solution for the in Patients With Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FE999306 CS01
Record Dates: First submitted 2011-11-16; First posted 2011-11-18 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Glycerol; Dioctyl Sulfosuccinic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docusate sodium and sorbitol rectal solution (Experimental)
  Interventions: Drug: Docusate sodium and sorbitol rectal solution
- Glycerine (Active Comparator)
  Interventions: Drug: Glycerine

INTERVENTIONS:
Drug: Glycerine
  Arms: Glycerine
Drug: Docusate sodium and sorbitol rectal solution
  Arms: Docusate sodium and sorbitol rectal solution

SUMMARY:
This study aims to evaluate the efficacy and safety of the docusate sodium and sorbitol rectal solution produced by Ferring Pharmaceutical (China) Ltd. in treating Chinese patients with constipation.

ELIGIBILITY:
Inclusion Criteria:

* Have signed the informed consent form and have been verbally told of the details of the trial and treatment procedures
* Is a citizen of the People's Republic of China
* Males and females aged between 18 and 65 years inclusive
* A history of constipation symptoms for at least 6 months, with occurrence of two or more of the symptoms during the 3 months before screening:

  1. More than 1/4 of stool classifiable as Type I or Type II on the Bristol Stool Scale;
  2. Sensation of incomplete evacuation at least 1/4 of the time;
  3. Straining during defecation at least 1/4 of the time;
  4. Sensation of ano-rectal blockage or obstruction during defecation at least 1/4 of the time;
  5. Manual manoeuvres needed often to facilitate defecations (e.g. digital evacuation) at least 1/4 of the time;
  6. Fewer than 3 bowel movements per week
* No bowel movement within two days prior to randomisation

Exclusion Criteria:

* Patients who are suspected to have colorectal cancer;
* Patients showing signs of bleeding in the digestive tract or inflammatory bowel disease;
* Patients experiencing abdominal discomfort or intestinal blockage for which the cause has yet to be determined;
* Patients allergic to docusate or sorbitol;
* Patients allergic to glycerine;
* Those pregnant, breastfeeding, or with the intention of becoming pregnant, or fertile women who are not on effective birth control（i.e. an IUD (intrauterine device), oral contraceptives or other obstructive measures;
* Severe liver damage (ALT (alanine aminotransferase), AST (aspartate transaminase), TBIL (serum total bilirubin) more than 2 times the upper limit of normal)
* Kidney function impairment (Cr (creatinine clearance rate), BUN (blood urea nitrogen) more than 1.5 times the upper limit of normal)
* Patients who have participated in any other clinical trial during the last 3 months;
* Diabetics who are currently undergoing insulin treatment;
* Patients who are unable to suspend using treatments that affect the kinetics of the digestive system in the 5 days prior randomisation. Such treatments include prokinetic drugs, erythromycin analogues, laxatives, etc;
* Other patient factor(s) (e.g. medical history, concurrent illness(es), laboratory test result(s), etc.) at Screening that in the opinion of the investigator(s) would put the trial patient at excessive risk;
* Patients who are unable to act in a legal capacity, unable to meet or perform study requirements, or are known or suspected as unable to comply with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Overall efficacy rate of the enema in treating the symptoms of constipation | Up to 30 minutes

SECONDARY OUTCOMES:
Time from conclusion of enema administration to patient's first bowel movement | Up to 30 minutes
Amount of straining that occurs during bowel movement (normal/difficult) | Up to 30 minutes
Feeling of emptying of the rectum post bowel movement (complete/incomplete) | Up to 30 minutes
Stool form after enema treatment according to Bristol Stool Scale | Up to 30 minutes
Anal complaints (absent, anal itch, anal irritation or anal pain) | Up to 30 minutes
Abdominal pain (absent, mild, moderate, or severe) | Up to 30 minutes
Patient's overall assessment of using the enema to treat the symptoms of constipation | Up to 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (9):
- China (9):
  - Southern Medical University - Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiaotong University Medical School - Renji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiaotong University Medical School - Ruijin Hospital, Shanghai, Shanghai Municipality